CLINICAL TRIAL: NCT01419184
Title: A Randomized Study to Evaluate Comparative Effectiveness, Inpatient Resource Utilization, and Cost of Daptomycin vs. Vancomycin in the Treatment of Patients With Complicated Skin and Skin Structure Infections Due to Suspected or Documented Methicillin-resistant Staphylococcus Aureus (MRSA)
Brief Title: Daptomycin Versus Vancomycin in Participants With Skin Infections Due to MRSA
Acronym: DAPHEOR1006
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3009-015; DAP-HEOR-10-06 (Other: Cubist Study Number)
Record Dates: First submitted 2011-08-16; First posted 2011-08-18 (Estimated); Results first posted 2015-07-08 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Staphylococcal Skin Infections
Keywords: Complicated Skin and Skin Structure Infections (cSSSI); Methicillin-resistant Staphylococcus aureus (MRSA); Daptomycin; Vancomycin; Antibiotics
MeSH Terms: conditions — Staphylococcal Skin Infections | interventions — Daptomycin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daptomycin (Experimental): 4 milligrams per kilogram (mg/kg) daptomycin administered intravenously (IV) once a day until end of antibiotic therapy for complicated skin and skin structure infections (cSSSI) or until hospital discharge, whichever occurred first. Investigators treated participants according to their usual decision-making and discretion.
  Interventions: Drug: Daptomycin
- Vancomycin (Active Comparator): Vancomycin was reconstituted per the manufacturer's instructions and was dosed per investigator's discretion and was administered IV until end of antibiotic therapy for cSSSI or until hospital discharge, whichever occured first. Investigators treated participants according to their usual decision-making and discretion
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Daptomycin
  Other Names: Cubicin
  Arms: Daptomycin
Drug: Vancomycin
  Arms: Vancomycin

SUMMARY:
This was a real-world, prospective, open-label, multicenter study in which participants were randomized (1:1) to receive intravenous (IV) vancomycin or IV daptomycin. The purpose of this study is to compare infection-related hospital length of stay, along with a number of participant-reported outcomes, between participants with complicated skin and soft tissue infection treated with daptomycin and vancomycin.

DETAILED DESCRIPTION:
Eligible participants will be recruited within 24 hours of hospital admission for cSSSI due to suspected or documented Methicillin-resistant Staphylococcus Aureus (MRSA), and who are anticipated to require IV antibiotics effective against MRSA and at least 3 days of hospitalization for management of cSSSI. The primary objective is to compare infection-related hospital length of stay between participants treated with daptomycin and vancomycin. Secondary objectives were to compare participant reported outcomes (pain symptoms and Health Related Quality of Life), 30 day cSSSI-related hospital readmission rates, and cSSSI-related medical resource utilization and costs between participants treated with daptomycin and vancomycin.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Primary reason for hospitalization is skin and skin structure infection of a complicated nature (for example, cellulitis/erysipelas, major cutaneous abscess, or wound infection) that requires IV antibiotic treatment for an anticipated 3 to14 days and hospitalization for management

  1. Further defined as infections either involving deeper soft tissue or requiring significant surgical intervention or infections in which the participant has a significant underlying disease state that complicates the response to treatment
  2. Are suspected or documented to be caused by MRSA
  3. At least 3 of the following clinical signs and symptoms associated with the cSSSI:

  i. Pain; tenderness to palpation; ii. Elevated temperature (>37.5°Celsius [99.5° Farenheit] oral or >38° Celsius [100.2° Farenheit] rectal); iii. Elevated white blood count (WBC) >10,000/millimeters cubed (mm^3); iv. Swelling and/or induration; erythema; v. Purulent or seropurulent drainage or discharge
* Physician determination that vancomycin or daptomycin would be the initial treatment of choice for the cSSSI under study (or meets institutional criteria for use of vancomycin or daptomycin)
* Informed consent obtained and signed
* Less than 24 hours post hospital admission

Exclusion Criteria:

* Participants with known bacteremia, osteomyelitis, septic arthritis, or endocarditis
* Conditions where surgery (in and of itself) constitutes curative treatment of the infection (for example, amputation, incision and drainage)
* cSSSIs which can be managed with an oral antibiotic
* Participants where hospitalization is expected to be <48 hours
* Nosocomial infection
* Participants with necrotizing infections or concomitant gangrene
* Use of systemic antibacterial therapy for the infection for > 24 hours within 48 hours prior to the start of study drug unless (a) the infecting Gram-positive pathogen was resistant in vitro to the therapy or (b) the therapy was administered for 3 or more days with either worsening or no improvement in the infection
* Pathogens identified at study entry to be nonsusceptible to daptomycin or vancomycin
* Participants with neutropenia or compromised immune function (that is, severe neutropenia [absolute neutrophil count <500 cells per microliter (μL)] or is anticipated to develop severe neutropenia during the study period due to prior or planned therapy)
* Renal insufficiency (calculated creatinine clearance [CLcr] <30 milliliters per minute or on dialysis)
* Known to be allergic or intolerant to daptomycin or vancomycin
* Pregnant or nursing mothers
* Suspected implanted device or prosthetic as source of infection
* Is considered unlikely to comply with study procedures or to be available for follow-up contact

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-09-09 (Actual); Primary Completion 2012-09-01 (Actual); Study Completion 2012-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cubist Pharmaceuticals Medical Monitor Medical Monitor, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (26):
- United States (25):
  - Mobile, Alabama
  - Chula Vista, California
  - Escondido, California
  - La Mesa, California
  - Oceanside, California
  - Augusta, Georgia
  - Decatur, Georgia
  - Waterloo, Iowa
  - Topeka, Kansas
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Royal Oak, Michigan
  - Minneapolis, Minnesota
  - Las Vegas, Nevada
  - Albany, New York
  - East Meadow, New York
  - Mineola, New York
  - The Bronx, New York
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Toledo, Ohio
  - Rapid City, South Dakota
  - Austin, Texas
- Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Kauf TL, McKinnon P, Corey GR, Bedolla J, Riska PF, Sims M, Jauregui-Peredo L, Friedman B, Hoehns JD, Mercier RC, Garcia-Diaz J, Brenneman SK, Ng D, Lodise T. An open-label, pragmatic, randomized controlled clinical trial to evaluate the comparative effectiveness of daptomycin versus vancomycin for the treatment of complicated skin and skin structure infection. BMC Infect Dis. 2015 Nov 7;15:503. doi: 10.1186/s12879-015-1261-9. PMID 26547411

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant enrolled in the study but was lost to follow up prior to being randomized to either treatment arm (daptomycin or vancomycin). This participant did not receive study drug and was not included in further analysis. No further details are available for this participant.
Groups:
- Daptomycin: Daptomycin 4 milligrams per kilogram (mg/kg) was administered intravenously once a day until end of antibiotic therapy for complicated skin and skin structure infections (cSSSI) or until hospital discharge, whichever occurred first. Investigators treated participants according to their usual decision-making and discretion.
Period: Overall Study
Arm/Group | Daptomycin | Vancomycin
Started | 128 | 121
Received at Least 1 Dose of Study Drug | 118 | 106
Completed | 118 (6 participants did not complete the study due to no valid infection-related length of stay (IRLOS)) | 106 (13 participants did not complete the study due to no valid infection-related length of stay (IRLOS))
Not Completed | 10 | 15
Not completed — Site data not available | 3 | 2
Not completed — No IRLOS-No in-patient end date reported | 3 | 6
Not completed — No IRLOS-randomized, not treated | 2 | 4
Not completed — No IRLOS-non trial antibiotic used | 1 | 2
Not completed — No IRLOS-No adverse event treatment date | 0 | 1
Not completed — Participant randomized, not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is drawn from the subset of the entire sample of participants that received at least 1 dose of study drug and that had complete data for calculating the primary outcome, infection-related length of stay (IRLOS).
Groups:
- Daptomycin: Daptomycin 4 milligrams per kilogram (mg/kg) was administered intravenously once a day until end of antibiotic therapy for cSSSI or until hospital discharge, whichever occurred first. Investigators treated participants according to their usual decision-making and discretion.
- Vancomycin: Vancomycin was reconstituted per the manufacturer's instructions and was dosed and administered intravenously until end of antibiotic therapy for cSSSI or until hospital discharge, whichever occurred first. Investigators treated participants according to their usual decision-making and discretion.
- Total: Total of all reporting groups
Arm/Group | Daptomycin | Vancomycin | Total
Number analyzed (Participants) | 118 | 106 | 224
Age, Customized [Number; unit: participants]
  18-29 Years Old | 16 | 10 | 26
  30-39 Years Old | 22 | 17 | 39
  40-49 Years Old | 30 | 21 | 51
  50-59 Years Old | 26 | 32 | 58
  60-69 Years Old | 14 | 21 | 35
  70+ Years Old | 10 | 5 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 49 | 103
  Male | 64 | 57 | 121

OUTCOME MEASURES:

1. Primary Outcome: Infection-Related Hospital Length of Stay
Description: Infection Related Hospital Length of Stay (IRLOS) is defined as the number of hours of hospitalization associated with antibiotic treatment of the complicated skin and skin structure infections (cSSSI) beginning at initiation of study-antibiotic administration and ending at discontinuation of all antibiotic therapy for cSSSI or at hospital discharge (whichever occurred first). This included continued hospitalization for treatment of adverse events resulting from use of the study antibiotic or subsequent antimicrobial therapy. The mean number of hours for each treatment group is presented.
Time Frame: Baseline (Day 0) through the End of Hospital Stay (up to Day 14)
Population: The primary analytic sample (subset of the entire sample) comprised participants receiving at least 1 dose of study drug with complete data to calculate the primary outcome, IRLOS. As the end of the IRLOS depended upon the participant's course of treatment, no static set of items were answered to determine if a participant had complete data.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 118 | 106
Hours | 91.46 (57.81) | 93.23 (60.78)

2. Secondary Outcome: Mean Change From Baseline to Hospital Discharge in Pain According to the Brief Pain Inventory-Short Form (BPI-SF)
Description: Pain was measured as the amount of pain experienced "right now" by the participant using an 11-point numerical rating scale adapted from Brief Pain Inventory-Short Form (BPI-SF). Participants were asked to rate pain in his or her skin infection from 0 to 10, where 0 is no pain and 10 is pain as bad as he or she could imagine. Change from baseline to hospital discharge is presented; a negative value represents a decrease in pain.
Time Frame: Baseline (Day 0), End of Hospital Stay (up to Day 14)
Population: The primary analytic sample (subset of the entire sample) comprised participants receiving at least 1 dose of study drug with complete data to calculate the primary outcome, IRLOS. Participants also had evaluable BPI-SF data at baseline and at hospital discharge.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 105 | 98
units on a scale | -2.08 (3.13) | -2.54 (3.46)

3. Secondary Outcome: Mean Change From Baseline to Hospital Discharge in Participant-reported Health-related Quality of Life (HRQoL)
Description: Health-related quality of life (HRQoL) was measured using the EuroQol-5 Dimensions, 5 Level (EQ-5D-5L) multi-attribute questionnaire. The 5 dimensions measured were: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant's health state was expressed by a descriptive profile of a 5 digit number. The EQ-5D health states were converted into a single summary index (from 0 to 1, with 0 representing death, to 1 representing perfect health) by applying weights to each of the levels in each dimension. Change from baseline to hospital discharge is presented; positive values represent an increase in health utility.
Time Frame: Baseline (Day 0), End of Hospital Stay (up to Day 14)
Population: The primary analytic sample (subset of the entire sample) comprised participants receiving at least 1 dose of study drug with complete data to calculate the primary outcome, IRLOS. Participants also had evaluable EQ-5D data at baseline and at hospital discharge.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 105 | 98
units on a scale | 0.12 (0.20) | 0.18 (0.21)

4. Secondary Outcome: Participant Global Impression of Improvement (PGI-I) at Hospital Discharge
Description: PGI-I assessments of improvement were measured by asking participants: How is your skin infection today compared to how it was yesterday? Scores were calculated based on response to the single item, where 1 = improved a lot; 2 = improved moderately; 3 = improved a little; 4 = no change; 5 = worsened a little; 6 = worsened moderately; 7 = worsened a lot. Mean PGI-I scores are presented at hospital discharge; lower values represent greater improvement.
Time Frame: End of Hospital Stay (up to Day 14)
Population: The primary analytic sample (subset of the entire sample) comprised participants receiving at least 1 dose of study drug with complete data to calculate the primary outcome, IRLOS. Participants also had evaluable PGI-I data at hospital discharge.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 102 | 97
units on a scale | 2.05 (1.16) | 1.80 (0.94)

5. Secondary Outcome: 30-day cSSSI-related Hospital Readmission Rates
Description: Hospital readmission rates were defined as readmission to an inpatient hospital facility within 30 days of hospital discharge for management of cSSSI relapse or treatment of adverse events related to cSSSI treatment. It did not include all-cause readmissions (for completeness, all-cause readmissions are reported in the descriptive tables). Participants were asked if they had been readmitted to the hospital since their discharge and whether the admission was specifically for their skin infection. The number of participants who were re-hospitalized for skin infection or side effects due to skin infection medication within 30 days since the initial hospital discharge (Day 14) is presented.
Time Frame: End of Hospital Stay (up to Day 14) through 30 days post hospital discharge
Population: The primary analytic sample (subset of the entire sample) comprised participants receiving at least 1 dose of study drug with complete data to calculate the primary outcome, IRLOS.
Measure: Number; unit: participants
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 118 | 106
participants | 5 | 2

6. Secondary Outcome: cSSSI-related Medical Resource Utilization and Costs
Description: Direct medical costs were based on utilization of health resources. Unit cost data were obtained from sources external to the trial and assigned to corresponding medical resource utilization observed within the trial to estimate costs of care. cSSSI-related costs were reported from a societal perspective, and further broken down into a health care system perspective. The health care system perspective includes hospital and outpatient costs. The societal perspective includes the health care system perspective plus participant and caregiver time loss from work and participant and caregiver out-of-pocket expenses. Total cost (including both total inpatient and total post-discharge costs) per participant is presented.
Time Frame: Baseline (Day 0) through 30 days post hospital discharge
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: dollars (United States)
Arm/Group | Daptomycin | Vancomycin
Number analyzed (Participants) | 118 | 106
dollars (United States)
  Health Care System Perspective | 10441.30 (7952.40) | 9894.34 (6620.51)
  Societal Perspective | 11085.57 (8120.20) | 10397.24 (6827.55)

ADVERSE EVENTS:
Description: Only serious adverse events were collected for this study.
Arm/Group | Daptomycin | Vancomycin
Serious Adverse Events (participants affected / at risk) | 15/118 | 9/106
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Daptomycin (N=118) | Vancomycin (N=106)
Atrial Fibrillation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Lyme infection, Lyme disease (General disorders) | 1 (1) | 0 (0)
Allergic reaction (dermatologic) (Immune system disorders) | 0 (0) | 1 (1)
Osteomyelitis, Foot (Infections and infestations) | 0 (0) | 1 (1)
Worsening infection to left hand due to non-compliance (Infections and infestations) | 1 (1) | 0 (0)
Right prepatella bursitis with abscess, Bursitis infective (Infections and infestations) | 1 (1) | 0 (0)
Acute Viral Syndrome (Infections and infestations) | 0 (0) | 1 (1)
Bilat Lower Extrem Cellulitis, Cellulitis of legs (Infections and infestations) | 1 (1) | 0 (0)
Chest Wall infection status post right breast implant removal (Infections and infestations) | 1/54 (1) | 0/49 (0)
Clinical worsening of right below knee stump infection (Infections and infestations) | 0 (0) | 1 (1)
Left hallux osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis with septic arthritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Right Leg Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
altered mental status (Psychiatric disorders) | 0 (0) | 1 (1)
respiratory failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
red man syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
social admission for reassignment of nursing home (Social circumstances) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other